CLINICAL TRIAL: NCT02457507
Title: Vitamin B12 Supplement to Prevent Cognitive Decline
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Timothy Kwok, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DM-B12
Record Dates: First submitted 2015-05-22; First posted 2015-05-29 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Vitamin B12 (Experimental): Vitamin B12, 1mg, daily, 27 months
  Interventions: Dietary Supplement: Vitamin B12
- Placebo (Placebo Comparator): Placebo comparator
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin B12 — 2 tablets
  Arms: Vitamin B12
Dietary Supplement: Placebo — 2 tablets
  Arms: Placebo

SUMMARY:
Background: Older diabetic people are at greater risk of cognitive decline than non-diabetic people. Vitamin B12 deficiency in older people is associated with cognitive impairment and Alzheimer's disease. Vitamin B12 deficiency may therefore contribute to cognitive decline in older diabetic people.

Objective: To determine whether the correction of mild vitamin B12 deficiency in cognitively normal older diabetic people reduces the incidence of cognitive decline.

Design: randomized, double blind, placebo controlled trial Subject: Cognitively normal diabetic outpatients aged 70 years or older with plasma vitamin B12 150-300 pmol/L in medical and family medicine/ general outpatient clinics.

Procedure: After excluding those with clinical manifestations of vitamin B12 deficiency and without family member who can reliably inform on cognitive functioning (personal contact at least once a week), eligible patients will be invited to participate in this clinical trial. After obtaining written consent, research assistant (RA) will record demographic and clinical information from the subjects and perform neuropsychological tests - 1. Clinical dementia rating scale (CDR), 2. neurocognitive test battery (see below) 3. Chinese Mini mental state examination (MMSE), 4. Geriatric depression scale (GDS). Fasting blood will be taken for serum methylmalonic acid (MMA). Those with cognitive impairment and significant comorbidities will be excluded.

264 eligible subjects will be randomly assigned to take either two Vitamin B12 500 microgram or two identical looking placebo tablets once daily for 27 months.

All subjects or family caregivers are reviewed in the research clinic every 12 weeks in which the research assistant performs a pill count and dispenses the trial tablets. At 9 monthly intervals, the subjects will have neurocognitive test battery repeated at research clinic. CDR will be repeated at month 18 and 27. At month 9 and 27, fasting serum MMA and vitamin B12 will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* >/= 70 years old
* B12: 150 - 300 pmol/L
* Caregiver (personal contact at least once a week)

Exclusion Criteria:

* Dementia
* Peripheral neuropathy
* Anaemia (Hb<10 g/dl)
* Renal failure (creatinine > 150 µmol/L
* Stroke

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 271 (Actual)
Dates: Start 2011-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in Clinical Dementia Rating Scale (CDR) | Change from baseline in CDR at month 9, 18, 27

SECONDARY OUTCOMES:
Change in Neurocognitive test battery (NTB) score | Change from baseline in NTB score at month 9, 18, 27
  NTB including tests of executive funciton, psychomotor speed and memory
Change in serum homocysteine (µmol/L) | Change from baseline in serum homocysteine at month 9, 27

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Kwok T, Lee J, Ma RC, Wong SY, Kung K, Lam A, Ho CS, Lee V, Harrison J, Lam L. A randomized placebo controlled trial of vitamin B12 supplementation to prevent cognitive decline in older diabetic people with borderline low serum vitamin B12. Clin Nutr. 2017 Dec;36(6):1509-1515. doi: 10.1016/j.clnu.2016.10.018. Epub 2016 Oct 27. PMID 27823800